CLINICAL TRIAL: NCT03658460
Title: Immune Checkpoint Inhibitors in Advanced Non-Small Cell Lung Cancer and Discovery of New Biomarkers
Acronym: LimBio
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Andreas Carus, Principal Investigator, Aalborg University Hospital
Other Study IDs: AaUH ONK 08-2018
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Non-small-cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; Lung Neoplasm
Keywords: immunotherapy; immune checkpoint inhibitors; biomarkers; sequencing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Sequence Analysis, DNA; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blod
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: DNA sequencing — Targeted next generation sequencing and gene expression analysis with focus on immuno-oncology signatures
  Other Names: Gene expression analysis

SUMMARY:
Lung cancer patients have a poor prognosis and only around 20 % is alive after 5 years. However, for advanced non-small cell lung cancer immunotherapy has become a cornerstone of treatment.

Two immunotherapeutic drugs for lung cancer have been approved in the last two years. Immunotherapy blocks the capability of cancer cells to inactivate the patient´s immune system, thus re-enabling eradication of cancer cells. In clinical trials, immunotherapy has shown superior survival and less toxicity compared to standard chemotherapy.

Whether the patients are candidates for immunotherapy or not is currently based on an unprecise biomarker that poorly predicts the patients who may benefit from immunotherapy. Immunotherapy can cause severe adverse effects and is expensive. Consequently, novel biomarkers are urgently needed from a patient perspective as well as a socioeconomic perspective.

The objective of the project is to investigate changes in genes and other signals in tissue and blood samples from immunotherapy treated lung cancer patients. The investigators expect to identify new biomarkers that can predict with high precision, which patients may benefit from immunotherapy. On-treatment, the investigators also aim to identify biomarkers that predict the treatment response and reveal the underlying mechanisms when cancer cells become resistant to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy verified NSCLC
* ≥ 18 years
* WHO/ECOG performance status ≤ 2
* Measurable disease according to RECIST 1.1
* Candidate for immunotherapy treatment
* Understand and accept oral and written information
* Written informed consent

Exclusion Criteria:

* Candidate for surgical and/or oncological treatment with curative intention
* Other synchronous cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Around 100 patients with advanced NSCLC, who meet the inclusion criteria, are consecutively included in the study. The outpatient clinic at the Departments of Oncology, Aalborg University Hospital and Aarhus University Hospital recruit and include the patients. Patients are candidates to the LimBio protocol regardless of immunotherapy treatment line.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Predictive, prognostic and resistance signatures | Until progression or 1 year after immunotherapy start date
  Next Generation Sequencing and gene expression analysis with NanoString PanCancer IO 360 panel in tissue samples at baseline and 1) at progression or 2) one year after immunotherapy start and no progression.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Carus, MD, PhD, Principal Investigator — Dept. of oncology, Aalborg University Hospital
Locations (1):
- Dept. of Oncology, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No